CLINICAL TRIAL: NCT03564613
Title: DOLOMITE NEAT ID Network Study: A Prospective, Multi-site Observational Study to Define the Safety and Effectiveness of Dolutegravir Use in HIV Positive Pregnant Women
Brief Title: Study to Define Safety and Effectiveness of Dolutegravir (DTG) Use in Human Immunodeficiency Virus (HIV) Positive Pregnant Women
Status: Recruiting | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 208759
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: HIV; Dolutegravir; Europe; NEAT ID; pregnancy; Safety; Antiretroviral
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV positive pregnant women: Data from approximately 250 HIV positive pregnant women with exposure to DTG from potential investigational sites across Europe will be included.
  Interventions: Drug: DTG

INTERVENTIONS:
Drug: DTG — Subjects with DTG exposure during any trimester will be included

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of DTG use in HIV positive pregnant women. This is a 3-year multi-site prospective observational study. Approximately, 250 HIV positive pregnant women from potential European AIDS Treatment Network (NEAT ID) sites across Europe will be enrolled. The enrollment period will be over 2 years with a follow-up period of 1 year for outcomes. The data collected will be that obtained during routine standard of care assessments; and the subjects will not undergo any interventional study procedures.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive pregnant women aged 18 years and over on DTG
* With no maternal or birth outcomes yet
* Subjects are able and willing to provide written informed consent and comply with any safety reporting requirements.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — HIV positive pregnant women
Study Population: Approximately, 250 HIV positive pregnant women having exposure to DTG from potential NEAT ID investigational sites across Europe will be enrolled.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of female subjects with spontaneous abortion | Up to 1 year
  Spontaneous abortion is defined as death of a fetus or expulsion of the products of conception before 22 weeks gestation.
Number of female subjects with induced abortion | Up to 1 year
  Induced abortion is defined as voluntary termination of pregnancy before 22 weeks gestation.
Number of female subjects giving still births | Up to 1 year
  Still birth is defined as the death of a fetus occurring at 22 weeks of gestation or more, or for situations in which the gestational age is unavailable, a fetus weighing at least 500 grams.
Number of female subjects with multiple births | Up to 1 year
  Number of female subjects giving multiple births will be reported.
Number of female subjects with type of deliveries | Up to 1 year
  The different type of deliveries will be summarized.
Maternal viral load (VL) at delivery | Up to 1 year
  The maternal viral load at the time of delivery will be summarized.
Number of infants with birth defects | Up to 1 year
  Birth defects will be classified according to World Health Organization's International Classification of Diseases, Tenth Revision.
Gestational age | Up to 1 year
  Number of females with birth collected data for gestational age as a measure of birth defects will be reported.
Birth weight | Up to 1 year
  Number of females with birth collected data for birth weight as a measure of birth defects will be reported.
Number of female subjects giving premature births | Up to 1 year
  Premature birth is defined as birth of live infant at <32 weeks gestation
Number of female subjects giving live births | Up to 1 year
  Number of female subjects giving live births will be reported.
Infants with low birth weight | Up to 1 year
  Low birth weight is defined as birth weight of <2500 grams.
Appearance, Pulse, Grimace, Activity, Respiration (APGAR) score in infants | Up to 1 year
  APGAR score in infants as a measure of birth defects will be calculated.
HIV status of Infants | Up to 1 year
  Infant's HIV status as a measure of birth defects will be reported.

SECONDARY OUTCOMES:
Number of female subjects with drug related Adverse Events and Serious Adverse Events | Up to 1 year
  Number of females with all drug related Adverse Events and Serious Adverse Events will be reported. These will be categorized by trimester of initiation.
Rate of DTG discontinuation in pregnant women | Up to 1 year
  Number of pregnant females with discontinuation of DTG will be reported.
Number of participants who discontinued DTG | Up to 1 year
  Reasons for DTG discontinuation will be summarized. Number of participants who discontinued DTG will be reported.
Number of participants with VL at discontinuation | Up to 1 year
  VL at discontinuation will be summarized to assess suppression. Number of participants with VL at discontinuation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No